CLINICAL TRIAL: NCT04122352
Title: The Effects of Trigger Point Treatment on Pain and Functionality in Temporomandibular Joint Dysfunction
Brief Title: The Effects of Trigger Point Treatment in Temporomandibular Joint Dysfunction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Ebru Kaya Mutlu, PT, Associate Prof. Dr, PhD, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2019/81
Record Dates: First submitted 2019-10-01; First posted 2019-10-10 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Temporomandibular Joint Dysfunction
Keywords: temporomandibular joint; trigger points; myofascial pain syndrome
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myofascial Pain Syndromes | interventions — Acupressure; Exercise

STUDY DESIGN:
Intervention Model Description: Individuals included in the study were randomized into two groups ; Group 1 : Exercises + ischemic compression Group 2 : Exercises
  Rocabado's 6x6 jaw exercises are shown to be applied to both groups for 4 weeks. After 1 week, posture exercises are added to the exercise programs of the patients.
  In addition to the exercises, Group 1 is given a total of 4 sessions of trigger point treatment after the initial evaluation, 1 week later, 2 weeks later and 4 weeks later.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercises + ischemic compression group (Experimental): volunteer patients with temporomandibular joint dysfunction with trigger points
  Interventions: Other: Ischemic compression; Other: Exercises (Rocabodo's 6x6 exercises and posture exercises)
- Exercises group (Other): volunteer patients with temporomandibular joint dysfunction with trigger points
  Interventions: Other: Exercises (Rocabodo's 6x6 exercises and posture exercises)

INTERVENTIONS:
Other: Ischemic compression — Ischemic compression was performed 3 times ; after the initial evaluation, after the first week evaulation and after the second week evaulations.
  Arms: Exercises + ischemic compression group
Other: Exercises (Rocabodo's 6x6 exercises and posture exercises) — Rocabodo's 6x6 exercises exercise was shown to be administered for 4 weeks. After the first week evaluation, posture exercises are added to the exercise programs of the patients.

SUMMARY:
The aim of this study to investigate the effectiveness of trigger point treatments (ischemic compression) on pain intensity, chronic pain severity, range of motion(ROM), pain pressure threshold (PPT) and functionality on patient with temporomandibular joint dysfunction.(TMD)

DETAILED DESCRIPTION:
TMD is most common of pain and functional limitations of jaw. The ischemic compression and the exercises (Rocabado's 6x6 exercises and posture exercises) each relieve pain and increase funcitonality on TMD but which one has the more effect should be investigated.

The ROCABODO's 6x6 exercise program, which is a special for temporomandibular joint, includes repetitive movements that include patient education, patient self-care, lifestyle modifications, and recognizing which actions have the effect of increasing the symptoms of an individual's active participation. The repetitive movements relax the chewing muscles and reduce pain by helping the synovial fluid move along the joint surfaces, increasing circulation, removing joint nutrition, and removing the metabolites of articular cartilage.

Postural exercise is commonly used for pain/tension in neck or back, but can also be applied in the orofacial region, aiming to relief muscle symptoms such as pain, tension, stiffness, and tiredness ,by improving the position of the head or the mandibular. It is believed that wrong head position can cause muscle pain due to acceleration of muscle activity in the neck and jaw muscles, as well as postural reflex. Postural exercise includes head posture correction and myofascial release.

Ischemic compression, that is a frequently used manual pressure technique, is a pressure application that is applied with the thumb to the maximum tolerable pain point on the trigger points. With this application, the sense of pain signals reduce pain by inhibiting the sense of touch signals.

The aim of this study to investigate the effectiveness of trigger point treatments (ischemic compression) on pain intensity, chronic pain severity, ROM, PPT and functionality on patient with TMD. 42 patients were randomized into 2 groups : Group 2 (n:21) received only exercises (Rocabado's 6x6 exercises and posture exercises) as treatment, Group 1(n:21) received exercises (Rocabado's 6x6 exercises and posture exercises) and ischemic compression as treatment.The rest, activity and night pain in activity were assessed by visual analog scale, ROM assessed by a ruler and PPT assessed by a digital algometer at baseline (before treatment), after 1week treatment, after 2 week treatment and after 4 week treatment. Chronic pain severity were assessed by Graded Chronic Pain Scale version 2 and functionality were assessed by Jaw Function Limitation Scale-8 at baseline (before treatment) and after 4 week treatment. The efect size was calculated for the assessments used in the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of TMD according to the criteria of DC / TMD (Diagnostic Criteria for Temporomandibular Disorders)
* Detection of trigger point during palpation of masticatory muscles
* Volunteer to participate in the study

Exclusion Criteria:

* To have undergone TMJ or cervical surgery and have been treated from these regions in the last 3 months
* Presence of rheumatic disease including TMJ
* Patients with TMJ instability or fractures
* Cases with cognitive impairment
* Presence of chronic pain such as trigeminal neuralgia
* Cases who do not regularly participate in treatment are excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2019-12-07 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | The rest, activity and night pain in activity were assessed by VAS at before and after 1 week of treatment, before and after 2 weeks of treatment, before and after 4 weeks of treatment.
  Pain intensity was assessed using the VAS; each patient was asked the pain during the rest, activity and at night (on a 0-10 numerical pain rating scale with zero corresponding to no pain and 10 corresponding to terrible pain). The rest, activity and night pain in activity were assessed by VAS at before and after 1 week of treatment, before and after 2 weeks of treatment, before and after 4 weeks of treatment.

SECONDARY OUTCOMES:
Graded Chronic Pain Scale version 2 (GCPS v2) | Chronic pain severity was assessed by GCPS v2 at before and after 4 weeks of treatment.
  Chronic pain severity was assesed using the GCPS v2. Scores are calculated for 3 subscales: the characteristic pain intensity score, which ranges from 0-100, is calculated as the mean intensity ratings for reported current, worst, and average pain; the disability score, which ranges from 0-100, is calculated as the mean rating for difficulty performing daily, social, and work activities; and the disability points score, which ranges from 0-3, is derived from a combination of ranked categories of number of disability days and disability score. The 3 subscale scores are used to classify subjects into 1 of the 5 pain severity grades: grade 0 for no pain, grade I for low disability-low intensity, grade II for low disability-high intensity, grade III for high disability-moderately limiting, and grade IV for high disability-severely limiting. Chronic pain severity was assessed by GCPS v2 at before and after 4 weeks of treatment.
Jaw Range of Motions (ROM) | ROM were assessed by a ruler at before and after 1 week of treatment, before and after 2 week of treatment, before and after 4 week of treatment.
  Jaw ROM measurements of unassisted painless mouth opening, maximum unassisted opening, maximum assisted opening, right lateral excursion and left lateral excursion were taken using a ruler. ROM were assessed by a ruler at before treatment, 1 week after start of treatment, 2 week after start of treatment and 4 week after start of treatment.
Jaw Functional Limitation Scale-8 (JFLS-8) | The functionality was assessed by JFLS-8 at before and after 4 weeks of treatment.
  The functionality was assessed using JFLS-8. The JFLS-8 was developed as an 8-item global scale for overall functional limitation of the masticatory system. All items are evaluated between 0 and 10. (0: no restrictions, 10: maximum restrictions) JFLS-8 are calculated as the mean of the available items. The functionality was assessed by JFLS-8 at before and after 4 weeks of treatment.
Pain Pressure Threshold (PPT) | PPT was evaluated by a digital algometer at before and after 1 week of treatment, before and after 2 weeks of treatment, before and after 4 weeks of treatment.
  PPT was assessed using the digital algometer. Assessment was performed massater, temporalis, lateral of the temporomandibular joint, sternocleidomastoideus and trapezius. PPT was evaluated by a digital algometer at before and after 1 week of treatment, before and after 2 weeks of treatment, before and after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Olcay Şakar, Prof. Dr., Principal Investigator — Istanbul University; Hanifegül Taşkıran, Prof. Dr., Principal Investigator — IstanbulAydın
Locations (1):
- Istanbul Aydin University, Istanbul, Bakırköy / Florya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shaffer SM, Brismee JM, Sizer PS, Courtney CA. Temporomandibular disorders. Part 1: anatomy and examination/diagnosis. J Man Manip Ther. 2014 Feb;22(1):2-12. doi: 10.1179/2042618613Y.0000000060. PMID 24976743
- [Result] McNeely ML, Armijo Olivo S, Magee DJ. A systematic review of the effectiveness of physical therapy interventions for temporomandibular disorders. Phys Ther. 2006 May;86(5):710-25. PMID 16649894
- [Result] Mulet M, Decker KL, Look JO, Lenton PA, Schiffman EL. A randomized clinical trial assessing the efficacy of adding 6 x 6 exercises to self-care for the treatment of masticatory myofascial pain. J Orofac Pain. 2007 Fall;21(4):318-28. PMID 18018993
- [Result] Cagnie B, Dewitte V, Coppieters I, Van Oosterwijck J, Cools A, Danneels L. Effect of ischemic compression on trigger points in the neck and shoulder muscles in office workers: a cohort study. J Manipulative Physiol Ther. 2013 Oct;36(8):482-9. doi: 10.1016/j.jmpt.2013.07.001. Epub 2013 Aug 28. PMID 23993756
- [Result] Schiffman E, Ohrbach R, Truelove E, Look J, Anderson G, Goulet JP, List T, Svensson P, Gonzalez Y, Lobbezoo F, Michelotti A, Brooks SL, Ceusters W, Drangsholt M, Ettlin D, Gaul C, Goldberg LJ, Haythornthwaite JA, Hollender L, Jensen R, John MT, De Laat A, de Leeuw R, Maixner W, van der Meulen M, Murray GM, Nixdorf DR, Palla S, Petersson A, Pionchon P, Smith B, Visscher CM, Zakrzewska J, Dworkin SF; International RDC/TMD Consortium Network, International association for Dental Research; Orofacial Pain Special Interest Group, International Association for the Study of Pain. Diagnostic Criteria for Temporomandibular Disorders (DC/TMD) for Clinical and Research Applications: recommendations of the International RDC/TMD Consortium Network* and Orofacial Pain Special Interest Groupdagger. J Oral Facial Pain Headache. 2014 Winter;28(1):6-27. doi: 10.11607/jop.1151. PMID 24482784
- [Result] Shaffer SM, Brismee JM, Sizer PS, Courtney CA. Temporomandibular disorders. Part 2: conservative management. J Man Manip Ther. 2014 Feb;22(1):13-23. doi: 10.1179/2042618613Y.0000000061. PMID 24976744